CLINICAL TRIAL: NCT05886049
Title: A Phase 1b Study of Menin Inhibitor SNDX-5613 in Combination With Daunorubicin and Cytarabine in Newly Diagnosed Patients With Acute Myeloid Leukemia and NPM1 Mutated/FLT3 Wildtype or MLL/KMT2A Rearranged Disease.
Brief Title: Testing the Addition of an Anti-cancer Drug, SNDX-5613, to the Standard Chemotherapy Treatment (Daunorubicin and Cytarabine) for Newly Diagnosed Patients With Acute Myeloid Leukemia That Has Changes in NPM1 or MLL/KMT2A Gene
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2023-04141; NCI-2023-04141 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10596 (Other: Ohio State University Comprehensive Cancer Center LAO); 10596 (Other: CTEP); UM1CA186712 (NIH)
Record Dates: First submitted 2023-06-01; First posted 2023-06-02 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-12

CONDITIONS: Acute Myeloid Leukemia With KMT2A Rearrangement; Acute Myeloid Leukemia With NPM1 Mutation
MeSH Terms: interventions — Specimen Handling; Biopsy; Cytarabine; Daunorubicin; revumenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (revumenib, daunorubicin, cytarabine) (Experimental): See Detailed Description.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Drug: Cytarabine; Drug: Daunorubicin; Procedure: Multigated Acquisition Scan; Drug: Revumenib; Procedure: Transthoracic Echocardiography Test

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Aspiration — Undergo bone marrow aspiration and biopsy
Procedure: Bone Marrow Biopsy — Undergo bone marrow aspiration and biopsy
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Drug: Cytarabine — Given IV
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-Cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Drug: Daunorubicin — Given IV
  Other Names: Daunomycin; Daunorrubicina; DNR; Leukaemomycin C; Rubidomycin; Rubomycin C
Procedure: Multigated Acquisition Scan — Undergo MUGA
  Other Names: Blood Pool Scan; Equilibrium Radionuclide Angiography; Gated Blood Pool Imaging; Gated Heart Pool Scan; MUGA; MUGA Scan; Multi-Gated Acquisition Scan; Radionuclide Ventriculogram Scan; Radionuclide Ventriculography; RNV Scan; RNVG; SYMA Scanning; Synchronized Multigated Acquisition Scanning
Drug: Revumenib — Given PO
  Other Names: Menin-Mixed Lineage Leukemia Protein-Protein Interaction Inhibitor SNDX-5613; Menin-MLL Inhibitor SNDX-5613; Menin-MLL Interaction Inhibitor SNDX-5613; SNDX 5613; SNDX-5613; SNDX5613
Procedure: Transthoracic Echocardiography Test — Undergo transthoracic ECHO
  Other Names: TRANSTHORACIC ECHOCARDIOGRAPHY; TTE

SUMMARY:
This phase Ib trial tests the safety, side effects, and best dose of SNDX-5613 when given in combination with the standard chemotherapy treatment (daunorubicin and cytarabine) in treating patients with newly diagnosed acute myeloid leukemia that has changes in the NPM1 gene or MLL/KMT2A gene. SNDX-5613 blocks signals passed from one molecule to another inside cancer cells that are needed for cancer cell survival. Drugs used in chemotherapy, such as daunorubicin and cytarabine, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Adding SNDX-5613 to the standard chemotherapy treatment may be able to shrink or stabilize the cancer for longer than the standard chemotherapy treatment alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD), recommended phase 2 dose (RP2D), and safety of revumenib (SNDX-5613) combined with 7 + 3 induction in newly diagnosed, untreated, NPM1-mutated/FLT3-ITD wild type and NPM1-mutated/FLT3-TKD wild type or MLL(KMT2A)-rearranged, acute myeloid leukemia (AML) patients >= 18-75 years old who are candidates for intensive induction therapy.

II. To determine the maximum tolerated dose (MTD), recommended phase 2 dose (RP2D), and safety of SNDX-5613 combined with one cycle of consolidation with high dose cytarabine in newly diagnosed AML patients in complete response/complete response with incomplete count recovery (CR/Cri) after intensive induction therapy with 7+3 for NPM1-mutated/FLT3-ITD wild type and NPM1-mutated/FLT3-TKD wild type or MLL (KMT2A)-rearranged AML patients >= 18-75 years old who are candidates for intensive therapy.

SECONDARY OBJECTIVES:

I. Evaluate the pharmacokinetics of SNDX-5613 with this combination regimen and characterize clinically relevant drug-drug interactions with antifungal agents.

II. To determine the number of patients with CR/CRi out of the total number of patients treated at each dose level of this regimen.

EXPLORATORY OBJECTIVES:

I. Explore potential biomarker indicators of response and resistance in AML samples.

II. To determine the measurable residual disease negative (MRD) response (CR/Cri) and its relation to CR/Cri status out of the total number of patients treated at each dose level of this regimen.

III. Determine number of patients that undergo hematopoietic stem cell transplant (HSCT) out of the total number of patients treated at each dose level of this regimen.

IV. Assess changes in OATP1B and CYP3A plasma biomarkers during treatment with SNDX-5613 with or without antifungal agents.

V. Determine duration of response.

OUTLINE: This is a phase Ib, dose-escalation study of revumenib followed by a dose-expansion study.

INDUCTION: Patients receive revumenib orally (PO) every 12 hours (Q12h) on days 2-28, daunorubicin intravenously (IV) over 15 to 30 minutes on days 1-3, and cytarabine by continuous IV infusion (CIV) on days 1-7 in the absence of disease progression or unacceptable toxicity. Patients who achieve a response to Induction treatment continue to Consolidation treatment. Patients with persistent disease continue to Re-Induction treatment. Patients also undergo a transthoracic echocardiogram (ECHO) or multigated acquisition scan (MUGA) during screening, bone marrow aspiration and biopsy during screening and at the end of Induction, and collection of blood during screening, on days 2, 3, 15, and at the end of Induction.

RE-INDUCTION: Patients receive revumenib PO Q12h on days 2-28, daunorubicin IV over 15 to 30 minutes on days 1-2, and cytarabine CIV on days 1-5 in the absence of disease progression or unacceptable toxicity. Patients who achieve a response to Re-Induction treatment continue to Consolidation. Patients also undergo a transthoracic ECHO or MUGA on day 1 and bone marrow aspiration and biopsy at the end of Re-Induction.

CONSOLIDATION: Patients receive revumenib PO Q12h on days 2-28 and cytarabine CIV on days 1-3 in the absence of disease progression or unacceptable toxicity. Patients also undergo bone marrow aspiration and biopsy at the end of Consolidation, and collection of blood on days 2, 3, 15, and at the end of Consolidation.

After completion of study treatment, patients are followed for 30 days or until death, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* Induction therapy: Patients ages 18-75 years at time of diagnosis with NPM1-mutated/FLT3-ITD wildtype and NPM1-mutated/FLT3-TKD wildtype or MLL (KMT2A) rearranged untreated AML and who are candidates for intensive induction chemotherapy
* Because no dosing or adverse event data are currently available on the use of SNDX-5613 in combination with daunorubicin and cytarabine in patients < 18 years of age, children are excluded from this study
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Total bilirubin =< 2 x institutional upper limit of normal (ULN), except for patients with Gilbert's syndrome
* Aspartate aminotransferase (AST)(serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT)(serum glutamic pyruvate transaminase [SGPT]) =< 3 x institutional upper limit of normal (ULN)
* Glomerular filtration rate (GFR) >= 60 mL/min/1.73 m^2 (via the Chronic Kidney Disease Epidemiology [CKD-EPI] glomerular filtration rate estimation)
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better
* Ejection fraction >= 50% (or >= 45% if no evidence of congestive heart failure [CHF] or other cardiac symptoms) by transthoracic echocardiogram (TTE) or multi-gated acquisition (MUGA) scan
* White blood cells (WBC) must be < 25 x 10^9/L. Hydroxyurea and leukapheresis are permitted to control the WBC prior to enrollment and initiation of protocol-defined therapy but must be stopped within 24 hours of initiation of protocol therapy. Must not have had any signs of leukostasis requiring cytoreduction
* Female patients of childbearing potential must agree to use 2 forms of contraception from screening visit until 120 days following the last dose of study treatment. Male patients of childbearing potential having intercourse with females of childbearing potential must agree to abstain from heterosexual intercourse or have their partner use 2 forms of contraception from screening visit until 120 days until the last dose of study treatment. They must also refrain from sperm donation from screening visit until 120 days following the last dose of study treatment
* Patients must have previously untreated AML with no prior treatment other than hydroxyurea. No chemotherapy for AML outside of hydroxyurea for treatment of leukostasis or all-trans retinoic acid (ATRA) for initially suspected acute promyelocytic leukemia (APL) (that is ruled out) is allowed
* Ability to understand and the willingness to sign a written informed consent document. Legally authorized representatives may sign and give informed consent on behalf of study participants

Exclusion Criteria:

* History of allergic reactions attributed to compounds of similar chemical or biologic composition to SNDX-5613, daunorubicin or cytarabine
* Patients with uncontrolled intercurrent illness that would make participation in this study unduly burdensome or unsafe for patient
* Patient must not have received known strong or moderate CYP3A4 inhibitors, or strong CYP3A4 inducers (with the exception of the antifungal) or sensitive/narrow therapeutic substrates of MATE1 within 7 days of enrollment. As part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product
* Pregnant women are excluded from this study because SNDX-5613 is a menin-KMT2A inhibitor agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with SNDX-5613, breastfeeding should be discontinued if the mother is treated with SNDX-5613. These potential risks may also apply to other agents used in this study
* Isolated myeloid sarcoma (i.e., patients must have blood or marrow involvement with AML to enter the study)
* Acute promyelocytic leukemia (French-American-British [FAB] M3)
* Active central nervous system (CNS) involvement by AML
* Uncontrolled symptomatic disseminated intravascular coagulopathy with active bleeding or signs of thrombosis
* Patients with Fridericia's correction formula (QTcF) >= 450 ms at screening; patients with right, left, or partial bundle branch blocks or a pacemaker who are asymptomatic are eligible regardless of QTC if cleared by cardiology for enrollment in the trial. Any factors that increase the risk of QTc prolongation or risk of arrhythmic event such as congenital long QT syndrome or family history of long QT syndrome
* Patients who will exceed a lifetime anthracycline exposure of > 550 mg/m^2 daunorubicin or equivalent (or > 400 mg/m^2 daunorubicin or equivalent in the event of prior mediastinal radiation) if they receive the maximum potential exposure to anthracyclines per protocol (including both induction and reinduction cycles)
* Patients with any gastrointestinal issue of the upper gastrointestinal (GI) tract that might affect oral drug absorption or ingestion (eg, gastric bypass, gastroparesis, etc)
* Patients who have cirrhosis with a Child-Pugh score of B or C
* Patients with Down Syndrome due to higher rates of chemotherapy-associated toxicities, and may have different pharmacokinetics, as well. Toxicities that occur at higher frequencies include cardiotoxicity, a known risk of SNDX-5613 treatment (i.e., QTcF prolongation)
* Patients with myelodysplastic syndromes (MDS) treated with previous intensive induction regimens similar to 7+3

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2024-06-20 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) for Induction | From day 1 to 42 of Induction or Re-Induction
  MTD of induction will be determined based on isotonic regression. Specifically, the MTD is selected as the dose for which the isotonic estimate of the toxicity rate is closest to the targeted dose-limiting toxicity (DLT) (i.e., 25%) via Bayesian Optimal Interval ("BOIN") software (MD Anderson). For all patients who receive at least one dose of any of the study drug(s), adverse events will be documented and summarized by type, grade, severity, and attribution using the Common Terminology Criteria for Adverse Events (CTCAE) version (v)5.0 criteria. In addition, the number of treatment cycles received and reasons for going off treatment will be summarized to assess treatment tolerability.
Maximum tolerated dose (MTD) for Consolidation | From day 1 to 42 of Consolidation
  MTD of induction will be determined based on isotonic regression. Specifically, the MTD is selected as the dose for which the isotonic estimate of the toxicity rate is closest to the targeted DLT (i.e., 25%) via "BOIN" software (MD Anderson). For all patients who receive at least one dose of any of the study drug(s), adverse events will be documented and summarized by type, grade, severity, and attribution using the CTCAE v5.0 criteria. In addition, the number of treatment cycles received and reasons for going off treatment will be summarized to assess treatment tolerability.
Recommended phase 2 dose for expansion cohort | From day 1 of Induction to day 42 of Consolidation
  For all patients who receive at least one dose of any of the study drug(s), adverse events will be documented and summarized by type, grade, severity, and attribution using the CTCAE v5.0 criteria. In addition, the number of treatment cycles received and reasons for going off treatment will be summarized to assess treatment tolerability.

SECONDARY OUTCOMES:
Pharmacokinetics (PK) of revumenib (SNDX-5613) | Cycle 1, day 2 at pre-treatment, 0.5, 1.0, 2.0, 4.0, 8.0 hours (hr); Cycle 1 day 3 at 12 hr; cycle 1 day 15 at pre-treatment, 0.5, 1.0, 2.0, 4.0, and 8.0 hr
  The PK sampling is designed to enable estimation of individual PK parameters of SNDX-5613 using standard noncompartmental methods. The primary analysis will compare SNDX-5613 exposure (area under the curve from zero to infinity [AUCinf]) on day 2 (before strong antifungal agent administration starting on Day 4 after completion of anthracycline) and steady-state exposure (area under plasma concentration-time curve over dosing interval [AUCtau]) on day 15 (after administration of antifungal agent).
Complete response/complete response with incomplete count recovery (CR/Cri) rate | At the end of cycle 1 of consolidation
  Will be calculated by the the number of patients achieving CR/CRi response out of the total number of patients treated on both the dose-escalation and expansion portions with 95% exact binomial confidence interveral.

OTHER OUTCOMES:
Best response to Induction | From day 1 to 42 of Induction or Re-Induction
  Will be determined for each patient using 2017 European LeukemiaNet criteria. The number of patients achieving response out of the total number of patients treated at a dose level will be described. Swimmer plots will be utilized to visually display how response improves/changes over time.
Best response overall | Up to 30 days after completion of study treatment
  Will be determined for each patient using 2017 European LeukemiaNet criteria. The number of patients achieving response out of the total number of patients treated at a dose level will be described. Swimmer plots will be utilized to visually display how response improves/changes over time.
Minimal residual disease (MRD) negative status | From day 1 to 42 of Induction, Re-Induction, and Consolidation
  MRD negative status is defined as the following for each genomic subgroup: 1) NPM1mutated/FLT3 ITD and FLT3 TKD wildtype: negative NPM1 by polymerase chain reaction testing on bone marrow after cycle 1 of consolidation (or after induction if unable to receive consolidation) or 2) MLL (KMT2A) rearrangement: negative multi-parameter flow cytometry (flow cutoff 10-3) after induction chemotherapy. The number of patients with MRD negative status and the relationship to clinical response will be described at each time point of interest. Swimmer plots will be utilized to visually display how MRD status improves/changes over time.
Duration of response | From the first date of complete response with incomplete count recovery or complete response until relapse or death from any cause, whichever occurs first, assessed up to 30 days after completion of study treatment
  Median survival will be estimated with 95% confidence interval using Kaplan-Meier method. Swimmer plots will be utilized to visually display how response improves/changes over time.
Overall survival | From the date on treatment until the date of death from any cause, assessed up to 30 days after completion of study treatment
  Median survival will be estimated with 95% confidence interval using Kaplan-Meier method. Swimmer plots will be utilized to capture milestone events including relapse of disease and death for each patient within a given dose level.
Number of patients who undergo hematopoietic stem cell transplant (HSCT) out of the total number patients treated at each dose level | Up to 30 days after completion of study treatment
  Will be described. Swimmer plots will be utilized to capture receipt of HSCT for each patient within a given dose level.
Changes in OATP1B and CYP3A biomarkers | Baseline to cycle 1, day 2 at pre-treatment, 0.5, 1.0, 2.0, 4.0, 8.0 hours (hr); Cycle 1 day 3 at 12 hr; cycle 1 day 15 at pre-treatment, 0.5, 1.0, 2.0, 4.0, and 8.0 hr
  Assess changes in OATP1B and CYP3A plasma biomarkers during treatment with SNDX-5613 with or without antifungal agents.

CONTACTS AND LOCATIONS:
Overall Officials: Alice S Mims, Principal Investigator — Ohio State University Comprehensive Cancer Center LAO
Locations (22):
- United States (22):
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - UM Sylvester Comprehensive Cancer Center at Aventura, Aventura, Florida
  - UM Sylvester Comprehensive Cancer Center at Coral Gables, Coral Gables, Florida
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Plantation, Plantation, Florida
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - University of Kansas Clinical Research Center, Fairway, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - University of Kansas Hospital-Indian Creek Campus, Overland Park, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Cincinnati Cancer Center-West Chester, West Chester, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - University of Virginia Cancer Center, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: Yes
"NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page."
URL: https://grants.nih.gov/policy/sharing.htm